CLINICAL TRIAL: NCT01108900
Title: Non-Interventional, Prospective Study Of the Evaluation Of Patients Population With ED, Treated With Sildenafil
Brief Title: A Study Of The Evaluation Of Patients Opulation With Erectile Dysfunction, Treated With Sildenafil
Acronym: SURE
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481271
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction udenafil sildenafil treatment satisfaction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with erectile dysfunction (ED): 100 ED patients in the study that were switched to sildenafil after a previous treatment with udenafil proved ineffective and/or was poorly tolerated
  Interventions: Drug: sildenafil

INTERVENTIONS:
Drug: sildenafil — tables, 25,50,100 mg, on demand, 1 month

SUMMARY:
In the present study, it is planned to observe a population of 100 ED patients treated previously with udenafil and for whom their physician decided to switch them to sildenafil because of poor udenafil tolerance and/or poor efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged ≥ 18 years.
* Clinical diagnosis of erectile dysfunction supported by a total score of less than or equal to 21 according to Sexual Health Inventory-Male (SHI-M).
* Patients having a sexual partner throughout the study.
* Patients having been switched to sildenafil after a previous treatment with udenafil proved ineffective and/or was poorly tolerated. The evaluation of udenafil ineffectivness should be performed after attempt intercourse 2 times a week over the course of four weeks.

Exclusion Criteria:

* The patients for whom sildenafil is contraindicated according to the Local Product Document (LPD). (See appendix D)
* The patients for whom sexual activity is not indicated.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients, aged >18 years and having been switched to sildenafil after a previous treatment with udenafil proved ineffective and/or was poorly tolerated. The evaluation of udenafil ineffectivness should be performed after attempt intercourse 2 times a week over the course of four weeks.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To observe the treatment satisfaction of ED patients (sum of questions 13-14 IIEF) that were switched to sildenafil after a previous treatment with udenafil proved ineffective and/or was poorly tolerated. | 1 month

SECONDARY OUTCOMES:
To evaluate a change of scores of the IIEF (sum of questions 1-5 and 15) and the EHS. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481271&StudyName=A%20Study%20Of%20The%20Evaluation%20Of%20Patients%20opulation%20With%20Erectile%20Dysfunction%2C%20Treated%20With%20Sildenafil